CLINICAL TRIAL: NCT03950310
Title: Evaluation of Myocardial Salvage by Scintigraphy After Excimer Laser Coronary Angioplasty and Percutaneous Coronary Intervention With Biodegradable-polymer Platinum Chromium Everolimus-eluting Stent in the Patients With Anterior ST Elevation Myocardial Infarction
Brief Title: Laser Atherectomy for ST Elevation Myocardial Infarction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID19, primary PCI number reduced.
Sponsor: Tokai University (Other)
Responsible Party: Principal Investigator, Yuji Ikari, MD PhD, Tokai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LASTPASS
Record Dates: First submitted 2019-04-20; First posted 2019-05-15 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
Keywords: ELCA; STEMI; Myocardial Salvage
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Masking Description: Open -but assessors are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELCA (Experimental): On the antegrade delivery of the laser catheter after wiring, we used safe laser techniques and injected saline before and during the laser procedure at a 0.5 mm/sec catheter advancement rate. Whether to perform a retrograde laser method depended on each operator. After ablation by ELCA, patients undergo balloon dilation via standard techniques, and as appropriate, receive drug-eluting stent deployment.
  Interventions: Device: Excimer laser catheter
- non ELCA (No Intervention): In non ELCA group, the conventional PCI procedure, including thrombus aspiration, POBA, and stent implantation was performed. The indication for aspiration was at the discretion of the physician based on angiographic, intravascular ultrasound, or optical coherence tomography/Optical Frequency-Domain Imaging.

INTERVENTIONS:
Device: Excimer laser catheter — The excimer laser catheter is equipped with multiple optical fibers on the periphery of the guide wire lumen corresponding to 0.014 inch, which is used for the purpose of reperfusion of barrier site of coronary artery. The connector on the front side is connected with the CVX-300 laser generator, and the tip at the top contact directly with the lesion. The laser catheter consisting of multiple optical fibers transmits the energy in the ultraviolet region from the CVX300 laser generator to the blockage in the blood vessel. The ultraviolet energy is transmitted from the tip of laser catheter, transpires the fibrous, calcified and arteriosclerotic lesion by light, and enables reperfusion in the lesion. The laser catheter has appropriate hydrophilic coating and easily follows the inside of coronary artery.
  Arms: ELCA

SUMMARY:
The objectives of this study are to observe and examine prospectively whether excimer laser coronary angioplasty (ELCA) and percutaneous coronary intervention with biodegradable-polymer platinum chromium everolimus-eluting stent may improve the myocardial salvage in the patients with anterior ST elevation myocardial infarction (STEMI) using the myocardial scintigram (acute-phase I123-BMIPP and chronic-phase 99mTc-tetrofosmin), and to clarify the myocardial protective effect of excimer laser in the patients with anterior STEMI.

DETAILED DESCRIPTION:
The clinical result of catheter treatment in the patients with acute myocardial infarction in these several decades improved because of progress of early reperfusion therapy and stent treatment technique. However, the no-reflow phenomenon is still remaining as a problem, which is involved in a decrease in left ventricular function and worsening of prognosis. It is considered that the no-reflow phenomenon is induced by atherosclerotic and thrombotic emboli, endothelial dysfunction of capillary vessels, free radicals and cytokine. The treatment combining the peripheral protection and thrombus aspiration aiming at prevention of no-reflow is expected to reduce no-reflow and the infarct size and has been conducted on the patients with acute myocardial infarction. However, a lot of randomized studies have been conducted, so far, which do not lead to reduction of infarct size and improvement of survival rate, and the efficacy has not been demonstrated.

Some explanations have been suggested for this phenomenon:

1. The operation method of device is complicated, and it is difficult to acquire the treatment technique.
2. Giant thrombus and solid lesion could not be aspirated effectively.
3. A lot of randomized studies have not focused on the "patients with anterior descending lesion of thrombolysis in myocardial infarction (TIMI) grade 0/1, of which the time from onset to treatment is within 6 hours," considered to have the largest benefit of prevention of no-reflow.

In recent years in Japan, excimer laser coronary angioplasty (ELCA) has been used in the patients with acute coronary syndrome (ACS), and not only debulking of arteriosclerotic lesion but also thrombolytic effect have been reported. In the Camel trial and Utility of Laser for Transcatheter Atherectomy Multicenter Analysis around Naniwa (ULTRAMAN) registry, the efficacy and safety in ACS have been reported, but the infarct size has not been evaluated.

This time in this study, it is considered that verification whether or not ELCA is able to improve the myocardial salvage in anterior ST elevation myocardial infarction (STEMI) using myocardial scintigram (acute-phase BMIPP and chronic-phase TF) will provide the useful information helpful for selection of treatment to medical care staffs and patients for future patients suffering from ACS and will be able to contribute to further improvement of medical science and medical practice.

MRI will be performed twice at 5-9 days and at 6 months post index ST elevation myocardial infarction to assess myocardial damage and functional variables, which details will be described in the following outcome measurement section.

ELIGIBILITY:
Inclusion Criteria:

* Patients to whom PCI treatment for anterior STEMI is indicated [Main selection criteria]
* First-episode anterior STEMI patients within 6 hours of onset that satisfy electrocardiogram criteria
* Patients who are 21 years of age or older at the time of consent acquisition
* Patient who the patient himself agreed in writing

Exclusion Criteria:

* Patients presenting cardiac shock at the time of visit
* Patients whose target lesions are left main trunk, circumflex, right coronary artery, distal anterior descending branch
* Patients who have TIMI 2, 3 at the initial imaging
* Patients with a reference vessel diameter of 2.5 mm or less
* Patients determined to lack consent ability for mental or other reasons
* Patient who is judged inappropriate by research researcher or research sharing doctor

The inclusion and exclusion criteria for the MRI will follow the main study, but in addition, will exclude following conditions.

* Atrial fibrillation subject at the timing of MRI scan
* Internally implanted devices such as pacemakers or ICDs
* Subject that is allergic to Gadolinium,
* Subject with claustrophobia
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
myocardial salvage (17 segment model) by SPECT | 3 day to 6 month
  Calculation of score using software in the Core Lab (Tokai University, Department of Radiology). Scoring should be conducted in 17 segments and at 5 grades from 0 to 4 in each segment on the polar map images. The Myocardial salvage (17-segment) was calculated by subtracting the total sum of the 123I-BMIPP and 99mTc-tetrofosmin defect scores in each segment ( ∑123I-BMIPP defect score minus 99mTc-∑tetrofosmin defect score).
Myocardial Salvage index (17 segment model) by SPECT | 3 day to 6 month
  Salvage index was calculated as follows: Myocardial Salvage index =∑123I-BMIPP defect score minus ∑99mTc-tetrofosmin defect score/ ∑123I-BMIPP defect score × 100 (%).

SECONDARY OUTCOMES:
Myocardial scar amount assessment by MRI | 5-9 days and 6 month
  All the outcome values will be derived by MRI image assessment. Each variables values will be derived as follows: Myocardial scar amount assessed on Late Short Axis LGE image
Microvascular obstruction assessment by MRI | 5-9 days and 6 month
  All the outcome values will be derived by MRI image assessment. Each variables values will be derived as follows: Microvascular obstruction on perfusion image and Early Short Axis LGE image
Myocardial salvage assessment by MRI | 5-9 days and 6 month
  All the outcome values will be derived by MRI image assessment. Each variables values will be derived as follows: Myocardial salvage derived from T2WBB and Late Short Axis LGE images
Ejection fraction assessment by MRI | 5-9 days and 6 month
  All the outcome values will be derived by MRI image assessment. Each variables values will be derived as follows: Ejection Fraction derived from Cine images
Gray zone assessment by MRI | 5-9 days and 6 month
  All the outcome values will be derived by MRI image assessment. Each variables values will be derived as follows: Gray zone derived from Late Short Axis LGE images.
Left ventricular ejection fraction by TF scintigraphy at 6 months | 5-7 month
  99mTc-tetrofosmin (TF) scintigraphy was performed 6 months after the PCI procedure. For the scanning procedure, the 740 MBq of 99mTc-tetrofosmin injected with patient while at rest. ejection fraction (%) based on 99mTc-tetrofosmin QGS data.
Left ventricular volume (ml) by TF scintigraphy at 6 months | 5-7 month
  99mTc-tetrofosmin (TF) scintigraphy was performed 6 months after the PCI procedure. For the scanning procedure, the 740 MBq of 99mTc-tetrofosmin injected with patient while at rest. Left ventricular volume (ml) based on 99mTc-tetrofosmin QGS data.
Left ventricular end-diastolic volume (ml) by TF scintigraphy at 6 months | 5-7 month
  99mTc-tetrofosmin (TF) scintigraphy was performed 6 months after the PCI procedure. For the scanning procedure, the 740 MBq of 99mTc-tetrofosmin injected with patient while at rest. Left ventricular end-diastolic volume (ml) based on 99mTc-tetrofosmin QGS data.
Left ventricular end-systolic volume (ml) by TF scintigraphy at 6 months | 5-7 month
  99mTc-tetrofosmin (TF) scintigraphy was performed 6 months after the PCI procedure. For the scanning procedure, the 740 MBq of 99mTc-tetrofosmin injected with patient while at rest. Left ventricular end-systolic volume (ml) on 99mTc-tetrofosmin QGS data.
Intra-stent tissue volume by OCT | at the end of procedure and 1-year
  OCT analysis should be conducted by an independent core lab (Kobe University Hospital) before and after stenting at Primary PCI and 1 year after PCI in selected patients. Should be conducted preoperatively, postoperatively and 1 year after operation. For analysis, the required matters (catheter size and target lesion) should be entered into the technician worksheet. The size and length of the stent used should be entered, in particular. In conducting OCI imaging in each medical institution, attention should be paid to the following points, and the requirements should be entered in the given section of technician worksheet: Analysis should be conducted based on the stent length described in the technician worksheet. In the qualitative analysis, the inside of stent and 5 mm to proximal and distal ends of stent should be evaluated at the interval of 0.2 mm. In the quantitative analysis, the inside of stent should be evaluated at the interval of 1.0 mm.
Myocardial salvage [total perfusion defect (TPD) model] by SPECT | 3 day to 6 month
  Myocardial salvage [total perfusion defect model (TPD)] = (Risk at area: TPD measured by BMIPP 3-9 days after p-PCI) minus (Infarct size: TPD measured by Tc99m-tetrofosmin at 6 months after p-PCI)
Myocardial salvage index (%) [total perfusion defect (TPD) model] by SPECT | 3 day to 6 month
  Myocardial salvage index (%) [total perfusion defect model (TPD)] = myocardial salvage / Risk at area: TPD measured by BMIPP 3-9 days after p-PCI x 100
Major adverse cardiovascular events (MACE) at 12 months | 12 months
  Major adverse cardiovascular events (MACE) MACE were defined as all-cause death, myocardial infarction (MI), or target lesion revascularization (TLR).
Major adverse cardiovascular events (MACE) at 36 months | 36 months
  Major adverse cardiovascular events (MACE) MACE were defined as all-cause death, myocardial infarction (MI), or target lesion revascularization (TLR).
Major adverse cardiovascular events (MACE) at 60 months | 60 months
  Major adverse cardiovascular events (MACE) MACE were defined as all-cause death, myocardial infarction (MI), or target lesion revascularization (TLR).
Cardiac death at 12 months | 12 months
  Death was considered to be of cardiac origin unless obvious noncardiac causes could be identified.
Cardiac death at 36 months | 36 months
  Death was considered to be of cardiac origin unless obvious noncardiac causes could be identified.
Cardiac death at 60 months | 60 months
  Death was considered to be of cardiac origin unless obvious noncardiac causes could be identified.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokai University School of Medicine, Isehara, Kanagawa, Japan

REFERENCES:
- [Background] Giugliano RP, Braunwald E; TIMI Study Group. Selecting the best reperfusion strategy in ST-elevation myocardial infarction: it's all a matter of time. Circulation. 2003 Dec 9;108(23):2828-30. doi: 10.1161/01.CIR.0000106684.71725.98. No abstract available. PMID 14662688
- [Background] Tanaka A, Kawarabayashi T, Nishibori Y, Sano T, Nishida Y, Fukuda D, Shimada K, Yoshikawa J. No-reflow phenomenon and lesion morphology in patients with acute myocardial infarction. Circulation. 2002 May 7;105(18):2148-52. doi: 10.1161/01.cir.0000015697.59592.07. PMID 11994247
- [Background] Gupta S, Gupta MM. No reflow phenomenon in percutaneous coronary interventions in ST-segment elevation myocardial infarction. Indian Heart J. 2016 Jul-Aug;68(4):539-51. doi: 10.1016/j.ihj.2016.04.006. Epub 2016 Apr 19. PMID 27543480
- [Background] Morishima I, Sone T, Okumura K, Tsuboi H, Kondo J, Mukawa H, Matsui H, Toki Y, Ito T, Hayakawa T. Angiographic no-reflow phenomenon as a predictor of adverse long-term outcome in patients treated with percutaneous transluminal coronary angioplasty for first acute myocardial infarction. J Am Coll Cardiol. 2000 Oct;36(4):1202-9. doi: 10.1016/s0735-1097(00)00865-2. PMID 11028471
- [Background] Ito H, Maruyama A, Iwakura K, Takiuchi S, Masuyama T, Hori M, Higashino Y, Fujii K, Minamino T. Clinical implications of the 'no reflow' phenomenon. A predictor of complications and left ventricular remodeling in reperfused anterior wall myocardial infarction. Circulation. 1996 Jan 15;93(2):223-8. doi: 10.1161/01.cir.93.2.223. PMID 8548892
- [Background] De Luca G, Ernst N, Zijlstra F, van 't Hof AW, Hoorntje JC, Dambrink JH, Gosslink AT, de Boer MJ, Suryapranata H. Preprocedural TIMI flow and mortality in patients with acute myocardial infarction treated by primary angioplasty. J Am Coll Cardiol. 2004 Apr 21;43(8):1363-7. doi: 10.1016/j.jacc.2003.11.042. PMID 15093868
- [Background] Rezkalla SH, Kloner RA. No-reflow phenomenon. Circulation. 2002 Feb 5;105(5):656-62. doi: 10.1161/hc0502.102867. No abstract available. PMID 11827935
- [Background] Stone GW, Webb J, Cox DA, Brodie BR, Qureshi M, Kalynych A, Turco M, Schultheiss HP, Dulas D, Rutherford BD, Antoniucci D, Krucoff MW, Gibbons RJ, Jones D, Lansky AJ, Mehran R; Enhanced Myocardial Efficacy and Recovery by Aspiration of Liberated Debris (EMERALD) Investigators. Distal microcirculatory protection during percutaneous coronary intervention in acute ST-segment elevation myocardial infarction: a randomized controlled trial. JAMA. 2005 Mar 2;293(9):1063-72. doi: 10.1001/jama.293.9.1063. PMID 15741528
- [Background] Ikari Y, Sakurada M, Kozuma K, Kawano S, Katsuki T, Kimura K, Suzuki T, Yamashita T, Takizawa A, Misumi K, Hashimoto H, Isshiki T; VAMPIRE Investigators. Upfront thrombus aspiration in primary coronary intervention for patients with ST-segment elevation acute myocardial infarction: report of the VAMPIRE (VAcuuM asPIration thrombus REmoval) trial. JACC Cardiovasc Interv. 2008 Aug;1(4):424-31. doi: 10.1016/j.jcin.2008.06.004. PMID 19463340
- [Background] Vlaar PJ, Svilaas T, van der Horst IC, Diercks GF, Fokkema ML, de Smet BJ, van den Heuvel AF, Anthonio RL, Jessurun GA, Tan ES, Suurmeijer AJ, Zijlstra F. Cardiac death and reinfarction after 1 year in the Thrombus Aspiration during Percutaneous coronary intervention in Acute myocardial infarction Study (TAPAS): a 1-year follow-up study. Lancet. 2008 Jun 7;371(9628):1915-20. doi: 10.1016/S0140-6736(08)60833-8. PMID 18539223
- [Background] Jolly SS, Cairns JA, Yusuf S, Meeks B, Pogue J, Rokoss MJ, Kedev S, Thabane L, Stankovic G, Moreno R, Gershlick A, Chowdhary S, Lavi S, Niemela K, Steg PG, Bernat I, Xu Y, Cantor WJ, Overgaard CB, Naber CK, Cheema AN, Welsh RC, Bertrand OF, Avezum A, Bhindi R, Pancholy S, Rao SV, Natarajan MK, ten Berg JM, Shestakovska O, Gao P, Widimsky P, Dzavik V; TOTAL Investigators. Randomized trial of primary PCI with or without routine manual thrombectomy. N Engl J Med. 2015 Apr 9;372(15):1389-98. doi: 10.1056/NEJMoa1415098. Epub 2015 Mar 16. PMID 25853743
- [Background] Frobert O, Lagerqvist B, Olivecrona GK, Omerovic E, Gudnason T, Maeng M, Aasa M, Angeras O, Calais F, Danielewicz M, Erlinge D, Hellsten L, Jensen U, Johansson AC, Karegren A, Nilsson J, Robertson L, Sandhall L, Sjogren I, Ostlund O, Harnek J, James SK; TASTE Trial. Thrombus aspiration during ST-segment elevation myocardial infarction. N Engl J Med. 2013 Oct 24;369(17):1587-97. doi: 10.1056/NEJMoa1308789. Epub 2013 Aug 31. PMID 23991656
- [Background] Stone GW, Dixon SR, Grines CL, Cox DA, Webb JG, Brodie BR, Griffin JJ, Martin JL, Fahy M, Mehran R, Miller TD, Gibbons RJ, O'Neill WW. Predictors of infarct size after primary coronary angioplasty in acute myocardial infarction from pooled analysis from four contemporary trials. Am J Cardiol. 2007 Nov 1;100(9):1370-5. doi: 10.1016/j.amjcard.2007.06.027. Epub 2007 Aug 17. PMID 17950792
- [Background] Nikolsky E, Stone GW, Lee E, Lansky AJ, Webb J, Cox DA, Brodie BR, Turco MA, Rutherford BD, Kalynych AM, Antoniucci D, Krucoff MW, Gibbons RJ, Fahy M, Mehran R. Correlations between epicardial flow, microvascular reperfusion, infarct size and clinical outcomes in patients with anterior versus non-anterior myocardial infarction treated with primary or rescue angioplasty: analysis from the EMERALD trial. EuroIntervention. 2009 Sep;5(4):417-24. doi: 10.4244/eijv5i4a66. PMID 19755327
- [Background] Topaz O, Minisi AJ, Bernardo NL, McPherson RA, Martin E, Carr SL, Carr ME Jr. Alterations of platelet aggregation kinetics with ultraviolet laser emission: the "stunned platelet" phenomenon. Thromb Haemost. 2001 Oct;86(4):1087-93. PMID 11686328
- [Background] Topaz O, Bernardo NL, Shah R, McQueen RH, Desai P, Janin Y, Lansky AJ, Carr ME. Effectiveness of excimer laser coronary angioplasty in acute myocardial infarction or in unstable angina pectoris. Am J Cardiol. 2001 Apr 1;87(7):849-55. doi: 10.1016/s0002-9149(00)01525-3. PMID 11274939
- [Background] Nishino M, Mori N, Takiuchi S, Shishikura D, Doi N, Kataoka T, Ishihara T, Kinoshita N; ULTRAMAN Registry investigators. Indications and outcomes of excimer laser coronary atherectomy: Efficacy and safety for thrombotic lesions-The ULTRAMAN registry. J Cardiol. 2017 Jan;69(1):314-319. doi: 10.1016/j.jjcc.2016.05.018. Epub 2016 Jul 2. PMID 27381939
- [Background] Rawlins J, Din JN, Talwar S, O'Kane P. Coronary Intervention with the Excimer Laser: Review of the Technology and Outcome Data. Interv Cardiol. 2016 May;11(1):27-32. doi: 10.15420/icr.2016:2:2. PMID 29588701
- [Derived] Kato Y, Lee WH, Natsumeda M, Ambale-Venkatesh B, Takagi K, Ikari Y, Lima JAC. Left atrial diastasis strain slope is a marker of hemodynamic recovery in post-ST elevation myocardial infarction: the Laser Atherectomy for STemi, Pci Analysis with Scintigraphy Study (LAST-PASS). Front Radiol. 2024 Feb 21;4:1294398. doi: 10.3389/fradi.2024.1294398. eCollection 2024. PMID 38450099